CLINICAL TRIAL: NCT04855851
Title: Effectiveness of Pain Neuroscience Education and Strength Training Program in Patients With Fibromyalgia
Brief Title: Effectiveness of Pain Neuroscience Education and Strength Training in Fibromyalgia
Acronym: PNE-ST-FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Rebollo Salas (Other)
Responsible Party: Sponsor-Investigator, Manuel Rebollo Salas, Director, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USeville-AJRD
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Education; Strength training
MeSH Terms: conditions — Fibromyalgia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAIN NEUROSCIENCE EDUCATION AND STRENGTH TRAINING (Experimental): Subjects will receive 6 PAIN NEUROSCIENCE EDUCATION (PNE) sessions and 12 weeks (3 times/week) of STRENGTH TRAINING (ST)
  Interventions: Procedure: PAIN NEUROSCIENCE EDUCATION AND STRENGTH TRAINING
- USUAL CARE (Active Comparator): The subjects of this group will receive Usual Care. In Spain, the treatment provided is mainly pharmacological, adjusted to the symptomatic profile of theses patients, and recommendation of aerobic and flexibility exercise
  Interventions: Procedure: USUAL CARE

INTERVENTIONS:
Procedure: PAIN NEUROSCIENCE EDUCATION AND STRENGTH TRAINING — The subjects of this group will receive an amount of six sessions that will be applied within 12 weeks. Every 15 days, the subjects will come for a consultation to receive a PNE session and review of the exercise program, which will be carried out 3 times a week for 12 weeks.
  Arms: PAIN NEUROSCIENCE EDUCATION AND STRENGTH TRAINING
Procedure: USUAL CARE — Aerobic exercises will consist of a standard table of low intensity stretching exercises, commonly prescribed to fibromyalgia patients. There will be three series of 30 seconds of each stretch, having a total duration of approximately 40 minutes. Each session will be held twice a week, following the recommendations of the "American College of Sport Medicine". Monitoring will be performed every 15 days by a physiotherapist.
  Arms: USUAL CARE

SUMMARY:
The main goal of this study is to get to know if applying both, pain neuroscience education (PNE) plus strength training (ST) will reduce the pain of fibromyalgia (FM). Both therapies have shown evidence of improvement in fibromyalgia patients. However, there are no studies evaluating their efficacy in combination.

DETAILED DESCRIPTION:
At present, the increase in knowledge about the neuroscience of pain has led to the integration of psychological factors, such as cognitions and beliefs about pain, fear-avoidance behaviors or catastrophism within the integrative perception of the concept . This has led to the development of therapeutic strategies aimed at the reconceptualization of pain through a treatment method called Pain Neuroscience Education (PNE), having shown evidence in the treatment of pain, disability, catastrophism and physical performance.

But despite current advances in pain neuroscience, there are still pain syndromes, such as fibromyalgia, that are the subject of debate and controversy. Fibromyalgia is a syndrome that causes generalized musculoskeletal pain, fatigue, sleep disorders, and physical disability. It is the main cause of chronic generalized musculoskeletal pain, with a prevalence of 1-5% of the world population. Scientific research has provided new insight for the diagnosis of fibromyalgia patients, who are characterized by a central sensitization process.

Objectives:

To assess the effectiveness of Pain Neuroscience Education and Strength Training to decrease pain and disability; and increasing quality of life and functionality in patients with Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with fibromyalgia.
* Duration of pain greater than one year.
* Generalized or present pain in more than two body regions.
* Not having participated in pain neuroscience education program.
* Not having participated in physical exercise programs in the last three months.

Exclusion Criteria:

* Presence of other diseases not related to the musculoskeletal system.
* Being under medical treatment not related to pain.
* being under physiotherapeutic treatment related to pain.
* Unavailability to carry out a physical exercise program.
* Pregnant or puerperium women.
* Inability to perform or complete the necessary tests to measure the study variables.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change from Self-report Pain Intensity | at the start of the study (at baseline, 0 week), after the last treatment session (12th week), 1 month from the last session (16th week), 3 months from the last session (20th week) and 6 months from the last session (32th week).
  Evaluated by the visual analogue scale (VAS). The total VAS score is between 0-10 cm. A higher score indicates greater pain intensity
Change from Central Sensitization symptoms | at the start of the study (at baseline, 0 week), after the last treatment session (12th week), 1 month from the last session (16th week), 3 months from the last session (20th week) and 6 months from the last session (32th week)
  Measured by the Central Sensitization Inventory (CSI). The total CSI score is between 0-100 points. Scores equal to or greater than 40 points are considered positive for Central Sensitization.
Change from Disability | at the start of the study (at baseline, 0 week), after the last treatment session (12th week), 1 month from the last session (16th week), 3 months from the last session (20th week) and 6 months from the last session (32th week)
  Measured by the Fibromyalgia Impact Questionnaire (FIQ). The total FIQ score is between 0-100. Thus, 0 represents the highest functional capacity and quality of life and 100 the worst state.

SECONDARY OUTCOMES:
Change from viscoelastic properties. | at the start of the study (at baseline, 0 week) and after 6 months from the last session (32th week)]
  Measured by the Myoton®.
Change from Autonomic Disfunction symptoms | at the start of the study (at baseline, 0 week) and after 6 months from the last session (32th week)]
  Measured by the Heart Rate Variability.
Change from Nerve Conduction Velocity | at the start of the study (at baseline, 0 week) and after 6 months from the last session (32th week)]
  Measured by the Sensory Nerve Action Potential (SNAP).
Change from grip strength | at the start of the study (at baseline, 0 week) and after 6 months from the last session (32th week)]
  Measure by the dynamometer.
Change from the pressure pain threshold | at the start of the study (at baseline, 0 week) and after 6 months from the last session (32th week)]
  Measure by the pressure algometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Investigación Área de Fisioterapia CTS 305 - Universidad de Sevilla, Seville, Spain, Spain

REFERENCES:
- [Background] Andrade A, de Azevedo Klumb Steffens R, Sieczkowska SM, Peyre Tartaruga LA, Torres Vilarino G. A systematic review of the effects of strength training in patients with fibromyalgia: clinical outcomes and design considerations. Adv Rheumatol. 2018 Oct 22;58(1):36. doi: 10.1186/s42358-018-0033-9. PMID 30657077
- [Background] Serrat M, Sanabria-Mazo JP, Garcia-Troiteiro E, Fontcuberta A, Mateo-Canedo C, Almirall M, Feliu-Soler A, Mendez-Ulrich JL, Sanz A, Luciano JV. Efficacy of a Multicomponent Intervention for Fibromyalgia Based on Pain Neuroscience Education, Exercise Therapy, Psychological Support, and Nature Exposure (NAT-FM): Study Protocol of a Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Jan 19;17(2):634. doi: 10.3390/ijerph17020634. PMID 31963773
- [Background] Nelson NL. Muscle strengthening activities and fibromyalgia: a review of pain and strength outcomes. J Bodyw Mov Ther. 2015 Apr;19(2):370-6. doi: 10.1016/j.jbmt.2014.08.007. Epub 2014 Aug 19. PMID 25892394
- [Background] Barrenengoa-Cuadra MJ, Angon-Puras LA, Moscosio-Cuevas JI, Gonzalez-Lama J, Fernandez-Luco M, Gracia-Ballarin R. [Effectiveness of pain neuroscience education in patients with fibromyalgia: Structured group intervention in Primary Care]. Aten Primaria. 2021 Jan;53(1):19-26. doi: 10.1016/j.aprim.2019.10.007. Epub 2020 Feb 6. Spanish. PMID 32033824
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Sarzi-Puttini P, Giorgi V, Marotto D, Atzeni F. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. Nat Rev Rheumatol. 2020 Nov;16(11):645-660. doi: 10.1038/s41584-020-00506-w. Epub 2020 Oct 6. PMID 33024295
- [Background] Marques AP, Santo ASDE, Berssaneti AA, Matsutani LA, Yuan SLK. Prevalence of fibromyalgia: literature review update. Rev Bras Reumatol Engl Ed. 2017 Jul-Aug;57(4):356-363. doi: 10.1016/j.rbre.2017.01.005. Epub 2017 Feb 8. English, Portuguese. PMID 28743363
- [Background] Cabo-Meseguer A, Cerda-Olmedo G, Trillo-Mata JL. Fibromyalgia: Prevalence, epidemiologic profiles and economic costs. Med Clin (Barc). 2017 Nov 22;149(10):441-448. doi: 10.1016/j.medcli.2017.06.008. Epub 2017 Jul 19. English, Spanish. PMID 28734619
- [Background] Yunus MB. Central sensitivity syndromes: a new paradigm and group nosology for fibromyalgia and overlapping conditions, and the related issue of disease versus illness. Semin Arthritis Rheum. 2008 Jun;37(6):339-52. doi: 10.1016/j.semarthrit.2007.09.003. Epub 2008 Jan 14. PMID 18191990
- [Background] Nijs J, Van Houdenhove B. From acute musculoskeletal pain to chronic widespread pain and fibromyalgia: application of pain neurophysiology in manual therapy practice. Man Ther. 2009 Feb;14(1):3-12. doi: 10.1016/j.math.2008.03.001. Epub 2008 Jun 3. PMID 18511329
- [Background] Cagnie B, Coppieters I, Denecker S, Six J, Danneels L, Meeus M. Central sensitization in fibromyalgia? A systematic review on structural and functional brain MRI. Semin Arthritis Rheum. 2014 Aug;44(1):68-75. doi: 10.1016/j.semarthrit.2014.01.001. Epub 2014 Jan 8. PMID 24508406
- [Background] Feliu-Soler A, Borras X, Penarrubia-Maria MT, Rozadilla-Sacanell A, D'Amico F, Moss-Morris R, Howard MA, Fayed N, Soriano-Mas C, Puebla-Guedea M, Serrano-Blanco A, Perez-Aranda A, Tuccillo R, Luciano JV. Cost-utility and biological underpinnings of Mindfulness-Based Stress Reduction (MBSR) versus a psychoeducational programme (FibroQoL) for fibromyalgia: a 12-month randomised controlled trial (EUDAIMON study). BMC Complement Altern Med. 2016 Feb 27;16:81. doi: 10.1186/s12906-016-1068-2. PMID 26921267
- [Background] Assumpcao A, Matsutani LA, Yuan SL, Santo AS, Sauer J, Mango P, Marques AP. Muscle stretching exercises and resistance training in fibromyalgia: which is better? A three-arm randomized controlled trial. Eur J Phys Rehabil Med. 2018 Oct;54(5):663-670. doi: 10.23736/S1973-9087.17.04876-6. Epub 2017 Nov 29. PMID 29185675
- [Background] American College of Sports Medicine Position Stand. The recommended quantity and quality of exercise for developing and maintaining cardiorespiratory and muscular fitness, and flexibility in healthy adults. Med Sci Sports Exerc. 1998 Jun;30(6):975-91. doi: 10.1097/00005768-199806000-00032. PMID 9624661
- [Derived] Rodriguez-Dominguez AJ, Rebollo-Salas M, Chillon-Martinez R, Cardellat-Gonzalez M, Blanco-Heras L, Jimenez-Rejano JJ. Pain Neuroscience Education and Resistance Training in Women With Fibromyalgia: A Randomized Control Pilot Study. Pain Res Manag. 2025 Jul 10;2025:7550108. doi: 10.1155/prm/7550108. eCollection 2025. PMID 40686548